CLINICAL TRIAL: NCT01146197
Title: Evaluation of Safety and Efficacity of Indometacin and Two Potassium Sparing Diuretics in Adult Patients Affected by Gitelman Syndrome
Brief Title: Input of the Use of Indometacin in Gitelman Syndrome as Compared to Potassium Sparing Diuretics
Acronym: GITAB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P071242
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Gitelman Syndrome
Keywords: Hypokalemia; Hypomagnesemia; Salt loosing nephropathy
MeSH Terms: conditions — Gitelman Syndrome; Hypokalemia | interventions — Therapeutics; Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Amiloride, Indometacin, Eplerenone (Experimental): Amiloride, indometacin(+Omeprazole), Eplerenone
  Interventions: Drug: TREATMENT
- Amiloride, Eplerenone, indometacin (Experimental): Amiloride, Eplerenone, indometacin (+Omeprazole)
  Interventions: Drug: TREATMENT
- Eplerenone, Amiloride, indometacin (Experimental): Eplerenone, Amiloride, indometacin (+Omeprazole)
  Interventions: Drug: TREATMENT
- Eplerenone, Indometacin, Amiloride (Experimental): Eplerenone, Indometacin, Amiloride
  Interventions: Drug: TREATMENT
- Indometacin, Eplerenone, Amiloride (Experimental): Indometacin, Eplerenone, Amiloride
  Interventions: Drug: TREATMENT
- Indometacin, Amiloride, Eplerenone (Experimental): Indometacin, Amiloride, Eplerenone
  Interventions: Drug: TREATMENT

INTERVENTIONS:
Drug: TREATMENT — Patients with received in random order 75mg/day indometacin(chronoindocid®), 10-20 mg/day amiloride and 50-150 mg /day eplerenone (Inspra ®). The three 6 weeks-periods of treatment will be followed by six weeks washout period. 3-6 weeks before the first period of treatment, a supplementation with potassium and magnesium will be orally given, and maintained at the same dose throughout the study and stoped 6 weeks after the end of the third period of treatment.
  Other Names: MODAMINE; Inspra and CHRONOINDOCID

SUMMARY:
Gitelman syndrome is a rare renal disease where the kidneys are unable to normally retain some salts (sodium, potassium and magnesium). Main consequences of these renal leaks of salts are a tendency toward low blood pressure, hypokalemia and hypomagnesemia both contributing to cardiac and muscles symptoms.

DETAILED DESCRIPTION:
Patients with received in random order 75mg/day indometacin (Chronoindocid®), 10-20 mg/day amiloride and 50-150 mg /day eplerenone (Inspra ®). The three 6 weeks-periods of treatment will be followed by six weeks washout period. 3-6 weeks before the first period of treatment, a supplementation with potassium and magnesium will be orally given, and maintained at the same dose throughout the study and stoped 6 weeks after the end of the third period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-60 yrs old, both sex, with genetically proven Gitelman's syndrome, under birth pill control for woman.

Exclusion Criteria:

* counter-indication to treatment under study
* Other diuretic or NAIS treatments than amiloride, spironolactone, or indometacin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of indomethacin on hypokalemia versus potassium and magnesium supplementation alone | 2 months

SECONDARY OUTCOMES:
To evaluate the effectiveness of indomethacin on disorders possibly induced by chronic hypokalemia and /or hypomagnesemia (EKG, lipid disorders related to insulin resistance, glucose/ insulin ratio) | 2 months
To evaluate the effectiveness of eplerenone and amiloride on hypokalemia. | 2 months
To evaluate and compare indomethacin, eplerenone or amiloride in terms of efficiency on biological and hormonal disorders | 2 months
  To evaluate and compare indomethacin, eplerenone or amiloride in terms of efficiency on biological and hormonal disorders other than hypokalemia (hypomagnesemia, hyperaldosteronism), glomerular filtration rate, hypotension, clinical tolerance, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Blanchard Anne, MD,PhD, Principal Investigator — APHP
Locations (1):
- Hopital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592